CLINICAL TRIAL: NCT05288218
Title: Evaluation of Leak-free Bronchoscope Adapter to Limit Ventilated Air Volume Loss and Pathogen Aerosolization From Intubated Patients Who Receive Bronchoscopy
Brief Title: Evaluation of Leak-free Bronchoscope Adapter
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling
Sponsor: Columbia University (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Beth Hochman, Assistant Professor of Surgery (in Anesthesiology), Dept of Surgery Acute Care, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAT3916
Record Dates: First submitted 2021-11-23; First posted 2022-03-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Insufficiency
Keywords: bronchoscopy; mechanical ventilation; hypoxemia; covid-19; pathogen spread
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; COVID-19

STUDY DESIGN:
Intervention Model Description: This study will compare the efficacy of the standard commercially available adapter to the newly developed leak-free adapter. The intervention is considered the "leak-free bronchoscope adapter." The study will be conducted as a randomized control trial in patients who require bronchoscopy. Once the participant has been randomized to either the "leak free adapter" vs. "standard adapter" group, the bronchoscope adapter will be spliced into the ventilator circuit. Bronchoscopy will then be performed by the primary critical care physician in the intensive care unit.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Leak-free bronchoscope adapter (Experimental): The mechanical ventilation circuit used in patients with respiratory failure is considered a closed-loop circuit between the patient and the ventilator. This allows air to flow from the ventilator to the patient and back to the circuit without escaping to the ambient environment. To perform bronchoscopy, a standard adapter is spliced into the ventilator circuit, which allows the bronchoscope to enter the ventilation circuit granting access to the patient's airways. This study will compare the efficacy of the standard commercially available adapter to the newly developed leak-free adapter. The intervention is considered the "leak-free bronchoscope adapter."
  Interventions: Device: Leak-free Bronchoscope Adapter
- Standard bronchoscope adapter (Active Comparator): The mechanical ventilation circuit used in patients with respiratory failure is considered a closed-loop circuit between the patient and the ventilator. This allows air to flow from the ventilator to the patient and back to the circuit without escaping to the ambient environment. To perform bronchoscopy, a standard adapter is spliced into the ventilator circuit, which allows the bronchoscope to enter the ventilation circuit granting access to the patient's airways. This study will compare the efficacy of the standard commercially available adapter to the newly developed leak-free adapter. This arm utilizes the standard adapter.
  Interventions: Device: Standard Bronchoscope Adapter

INTERVENTIONS:
Device: Leak-free Bronchoscope Adapter — A novel leak-free bronchoscope adapter will connect to the ventilation circuit in place of a standard adapter.
  Arms: Leak-free bronchoscope adapter
Device: Standard Bronchoscope Adapter — Commercially available bronchoscope adapter (Smiths Medical)
  Arms: Standard bronchoscope adapter

SUMMARY:
Patients who develop respiratory failure require the assistance of mechanical ventilation while recovering from their respiratory injury. For example, patients that are affected by COVID-19 can develop such severe respiratory failure that they are unable to breathe on their own and therefore require the assistance of a mechanical ventilator. A Bronchoscope is a tool that can be used to visualize the inside of the lungs to aid in further diagnosis and delivery of therapeutic agents in patients with respiratory disease or failure. However, bronchoscopy can cause air to leak from the patient's lungs into the room due to a poorly designed adapter that is required to facilitate the introduction of the bronchoscope into the lungs. This leak can lead to the patient losing oxygen during the procedure which can be harmful to the patient and delay or limit recovery. Additionally, the air that leaks can lead to the spread of bacteria/viruses into the ambient air, which can contaminate the intensive care unit and expose other patients and healthcare workers to harmful pathogens. This was highlighted most recently during the COVID-19 pandemic where national guidelines limited the use of bronchoscopy in patients affected by the virus due to concerns about spreading the virus within the hospital and to the healthcare workers.

In this study, the investigators will evaluate the efficacy of a novel adapter that avoids air leakage during bronchoscopy. Patients with respiratory failure on mechanical ventilation who require bronchoscopy will be randomized into two groups (groups A and B). These patients will be identified by the intensive care unit physician. Informed consent will be obtained from the patient's health care proxy. Patients in group A will undergo bronchoscopy using the standard commercially available adapter. Patients in group B will undergo bronchoscopy using the newly developed bronchoscope adapter. The efficacy of the bronchoscopy adapter will be evaluated by analyzing ventilator-associated parameters as well as the level of air contamination after the procedure. A bronchoscope adapter that limits air leak would have significant value in improving patient outcomes who receive bronchoscopy. Additionally, this would allow bronchoscopy to be more readily performed in patients with potential bacterial/viral pathogen spread.

Primary objective: Determination of equivalency or superiority of the new "leak-free adapter" compared to the standard commercial adapter to enable safe bronchoscopy in ventilated patients requiring bronchoscopy.

Secondary objective: To determine if the adapter provides improved ventilation during bronchoscopy by limiting tidal volume loss and pathogen aerosolization.

DETAILED DESCRIPTION:
Patients who develop acute respiratory failure require hospitalization and mechanical ventilatory support. Of all patients admitted to intensive care units in the US, approximately 40% require mechanical ventilation. With the ongoing COVID-19 pandemic, approximately 18% of affected patients are expected to require mechanical ventilation.

Mechanical ventilation requires endotracheal intubation (cannulation of the patient's trachea) to deliver ventilated air to the lungs. Air is delivered by the ventilator to the patient using positive pressure in a closed circuit, ensuring adequate tidal volume to the patient without air escape to the outside environment. Nevertheless, patients placed on mechanical ventilation often develop superimposed infections known as "Ventilator-Associated Pneumonia" (VAP) as well as significant mucus secretions which limit effective mechanical ventilation. A camera tipped device is used to enable more effective bronchoscopy to visualize and explore the tracheobronchial tree for both diagnostic (bacterial/viral sampling) and therapeutic (suctioning obstructive mucus secretions, delivery of therapeutic agents) purposes.

Despite clear diagnostic and therapeutic benefits, bronchoscopy is also associated with substantial morbidity and complications. To perform bronchoscopy, a standard (commercially available) adapter allows the bronchoscope to enter the closed ventilation circuit, providing direct access to the patient's airways. However, the standard adapter leads to a significant leak of tidal volume outside of the ventilation circuit to the ambient environment. This air leak from the adapter leads to two major complications: First, the loss of positive pressure ventilation to patients means that oxygen is not being delivered to the patient and therefore leads to hypoxemia, which limits the duration and efficacy of bronchoscopy. Second, escaped air from the ventilator circuit can lead to the generation of aerosols, which can lead to the significant spread of viral and bacterial infectious agents to the ambient environment and surrounding healthcare providers. Intensive care units (ICUs) in the US must employ negative pressure ventilation to limit pathogen spread outside of the room and to the rest of the ICU. ICU rooms equipped with standard room negative pressure ventilation require 46 minutes after bronchoscopy to clear 99% of aerosolized pathogens. Thus, despite the known diagnostic and therapeutic benefits of bronchoscopy, concerns surrounding viral exposure related to an air leak from bronchoscopy adapters led to the development of national guidelines that limited bronchoscopy in patients affected by Covid-19.

To overcome these limitations, the investigators developed a novel bronchoscope adapter capable of effectively limiting all tidal volume loss (i.e., air leak via adapter) associated with the currently available standard adapters. In ex-vivo and animal studies, the investigators noted that a significant portion of tidal volume delivered by the ventilator is lost to the ambient air when using the standard bronchoscope adapter using the standard adapter (~40%). There was no tidal volume loss associated with the Leak-free bronchoscope adapter. The innovation in this adapter's development lies in the capacity to form an improved seal around the bronchoscope that limits tidal volume loss around the bronchoscope and captures air that escapes the circuit with the insertion and removal of the bronchoscope. Of note, the adapter is positioned outside the circuit and is only a conduit for the bronchoscope to enter the circuit.

Here the investigators propose a comparative effectiveness study that evaluates the leak-free bronchoscope adapter's use to enable bronchoscopy similar to the standard adapter. Additionally, the investigators will evaluate the adapter's capacity to deliver either equivalent tidal volume to the currently available adapter in patients undergoing bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with respiratory failure who require mechanical ventilation for any reason except those listed below (exclusion criteria).
2. Male or female
3. Aged 18 years or above

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. Female participants who are pregnant during the study.
2. SpO2 (oxygen saturation) < 90% at baseline.
3. The patient requires high ventilation requirements as indicated by a positive end-expiratory pressure (PEEP) greater than 20 mmHg or inspired oxygen requirements greater than 90%.
4. Hemodynamic instability requiring significant use of vasoactive pressors to maintain blood pressure.
5. Any other significant disease or disorder that, in the Investigator's opinion, may either put the participants at risk because of participation in the study or may influence the result of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of tidal volume loss during procedure | Baseline and at one minute into the procedure
  To measure tidal volume loss, the patient's ventilator displays both total volume of inspired (VTi) air and expired (VTe) air for each breath given. Immediately prior to the start of bronchoscopy, baseline values for VTi and VTe will be recorded for 10 breaths. Upon initiation of bronchoscopy, the VTi and VTe values will be recorded for 10 breaths one minute after the initiation of the bronchoscopy procedure.
Change from baseline of oxygen saturation levels during procedure | Baseline and at one minute into the procedure
  To measure patient oxygen saturation (SpO2) as measured using a pulse oximeter through the procedure. Immediately prior to bronchoscopy, the patient's baseline circulating oxygen saturation will be recorded during 10 ventilated breaths. One minute after initiation of bronchoscopy, the SpO2 level will be recorded for 10 breaths during the procedure. The oxygen saturation sensor is a standard non-invasive device placed on the patient and provides continuous pulse oximetry monitoring.
Change from baseline of Particulate matter (PM) in air immediately post-procedure | Baseline and at one minute post-procedure
  Air quality samples will be obtained to monitor the level and degree of circulating particulate matter using an air quality sampler. The sampling device will obtain an air sample immediately before the bronchoscopic procedure as baseline, and a second sample will be obtained immediately after the procedure. The sampling device is a non-invasive tool placed within the room and near the participant during the procedure.
Change from baseline of aerosolized pathogens immediately post-procedure | Baseline and at one minute post-procedure
  Air quality samples will be obtained to monitor the level and degree of aerosolized pathogens using an air quality sampler. The sampling device will obtain an air sample immediately before the bronchoscopic procedure as baseline, and a second sample will be obtained immediately following the procedure. The sampling device is a non-invasive tool placed within the room and near the participant during the procedure.
Change from baseline of Pulmonary dynamic compliance immediately post-procedure | Baseline and at one minute post-procedure
  Immediately prior to initiating the bronchoscopic procedure, a baseline pulmonary dynamic compliance value will be obtained from the ventilator. The ventilator provides this continuous value in all intubated patients. A repeat value will then be obtained immediately following the completion of the bronchoscopic procedure.

SECONDARY OUTCOMES:
Change from baseline of Heart rate during procedure | Baseline and at one minute into the procedure
  Immediately prior to the initiation of the bronchoscopic procedure, the patient's baseline heart rate will be recorded. These values will be continuously monitored throughout the bronchoscopic procedure and recorded through the bronchoscopic procedure.
Change from baseline of systolic and diastolic blood pressure during procedure | Baseline and at one minute into the procedure
  Immediately prior to the initiation of the bronchoscopic procedure, the patient's baseline systolic and diastolic blood pressure will be recorded. These values will be continuously monitored throughout the bronchoscopic procedure and recorded through the bronchoscopic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Hochman, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No
Patient data is anonymized for study analysis. There are no plans to share data beyond the scope of researchers directly involved with this study.

REFERENCES:
- [Background] Wunsch H, Wagner J, Herlim M, Chong DH, Kramer AA, Halpern SD. ICU occupancy and mechanical ventilator use in the United States. Crit Care Med. 2013 Dec;41(12):2712-9. doi: 10.1097/CCM.0b013e318298a139. PMID 23963122
- [Background] Cummings MJ, Baldwin MR, Abrams D, Jacobson SD, Meyer BJ, Balough EM, Aaron JG, Claassen J, Rabbani LE, Hastie J, Hochman BR, Salazar-Schicchi J, Yip NH, Brodie D, O'Donnell MR. Epidemiology, clinical course, and outcomes of critically ill adults with COVID-19 in New York City: a prospective cohort study. Lancet. 2020 Jun 6;395(10239):1763-1770. doi: 10.1016/S0140-6736(20)31189-2. Epub 2020 May 19. PMID 32442528
- [Background] Kalanuria AA, Ziai W, Mirski M. Ventilator-associated pneumonia in the ICU. Crit Care. 2014 Mar 18;18(2):208. doi: 10.1186/cc13775. No abstract available. PMID 25029020
- [Background] Chhajed PN, Glanville AR. Management of hypoxemia during flexible bronchoscopy. Clin Chest Med. 2003 Sep;24(3):511-6. doi: 10.1016/s0272-5231(03)00050-9. PMID 14535223
- [Background] Tran K, Cimon K, Severn M, Pessoa-Silva CL, Conly J. Aerosol generating procedures and risk of transmission of acute respiratory infections to healthcare workers: a systematic review. PLoS One. 2012;7(4):e35797. doi: 10.1371/journal.pone.0035797. Epub 2012 Apr 26. PMID 22563403